CLINICAL TRIAL: NCT07204197
Title: Investigation of the Effectiveness of Virtual Reality-Assisted Physical Therapy in the Acute Period After Lumbar Disc Surgery
Brief Title: Effectiveness of Virtual Reality-Assisted Physical Therapy in the Acute Phase After Lumbar Disc Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assistant Professor, Department of Neurological Physiotherapy and Rehabilitation, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRLDHS1D
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Herniation; Lumbar Disc Surgery
Keywords: lumbar disc herniation; lumbar disc surgery; physiotherapy and rehabilitation; virtual reality; pain; functional capacity; psychosomatic status
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, controlled, parallel-group design. Participants undergoing lumbar disc surgery will be randomly assigned to one of two groups: (1) Virtual Reality-Assisted Physical Therapy or (2) Conventional Physical Therapy. Both groups will receive interventions starting from postoperative day 1, until the day of discharge and outcomes will be compared between the two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual-Reality-Assisted Physical Therapy Group (Experimental): Participants assigned to this group will receive a standardized 40-minute physical therapy program starting on postoperative day 1, followed by a 20-minute immersive virtual reality (VR) session. The VR application provides a relaxation-focused, interactive environment designed to reduce pain perception, anxiety, and stress while supporting engagement in rehabilitation. Sessions are delivered once daily during hospitalization. Patients are monitored for comfort and potential side effects such as dizziness or nausea, and all procedures are supervised by a physiotherapist to ensure safety and adherence.
  Interventions: Other: Virtual Reality-Assisted Physical Therapy
- Conventional Physical Therapy Group (Active Comparator): Participants in this group will receive the same standardized physical therapy program as the VR group, beginning on postoperative day 1. To match the 60-minute session length, exercise repetitions and intensity are increased instead of adding virtual reality. Thus, both groups complete identical physical therapy content, with the only difference being the addition of a VR session in the intervention group. All sessions are delivered once daily during hospitalization and supervised by a physiotherapist.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Virtual Reality-Assisted Physical Therapy — VR Assisted PT intervention, combines a standardized postoperative physical therapy program with an additional 20-minute immersive VR session. The VR component is relaxation-focused and interactive, making the total session length 60 minutes. The distinguishing feature is the integration of VR technology into early rehabilitation after lumbar disc surgery, which is not part of conventional therapy.
  Other Names: Conventional Physical Therapy
  Arms: Virtual-Reality-Assisted Physical Therapy Group
Other: Conventional Physical Therapy — This intervention consists of the same standardized physical therapy program as the VR group, delivered for 60 minutes daily by increasing exercise repetitions and intensity. The distinguishing feature is that it does not include any VR component, allowing direct comparison of physical therapy alone versus VR-assisted therapy.
  Arms: Conventional Physical Therapy Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of virtual reality-assisted physical therapy in the acute postoperative period after lumbar disc surgery.

The main questions it aims to answer are:

* Does virtual reality-assisted physical therapy reduce pain more effectively than conventional physical therapy?
* Does it improve functional recovery, pain threshold, and blood biomediator levels?
* Does it reduce anxiety and kinesiophobia in the early rehabilitation period?

Researchers will compare virtual reality-assisted physical therapy with standard physical therapy to determine whether virtual reality provides additional therapeutic benefits.

Participants will:

* Undergo standard postoperative physical therapy after lumbar disc surgery.
* Some participants will additionally perform virtual reality-based rehabilitation exercises.
* Be evaluated for pain severity, functional improvement, blood biomediators, pain threshold, and psychological outcomes.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is one of the most common musculoskeletal disorders and a major cause of low back pain worldwide. It occurs when the intervertebral disc extends beyond its anatomical boundaries, compressing neural structures and leading to pain, disability, and reduced quality of life. Although most patients are treated conservatively, approximately 15% require surgical intervention. Postoperative pain is one of the most significant challenges after lumbar disc surgery, reported in up to 70% of patients in the acute period. Insufficient pain management may delay mobilization, prolong hospitalization, increase healthcare costs, and negatively affect both physical and psychological recovery.

Pharmacological treatments, such as NSAIDs, opioids, muscle relaxants, and neuropathic pain agents, are commonly used for postoperative pain control. However, their potential side effects and limited efficacy have raised interest in non-pharmacological interventions. Conventional physical therapy protocols-mobilization, exercise, manual therapy, and patient education-are central to postoperative rehabilitation, improving mobility, functional recovery, and independence. Early mobilization within the first days after surgery has been shown to reduce complications and accelerate healing.

In recent years, technology-based approaches have emerged as complementary or alternative rehabilitation methods. Among them, virtual reality (VR) offers interactive, multisensory, and engaging environments that can contribute to both physical and psychological recovery. VR has shown therapeutic potential in pain management by diverting attention, reducing anxiety and stress, and promoting patient engagement in rehabilitation. Importantly, VR has demonstrated effectiveness in musculoskeletal conditions, neurological rehabilitation, and postoperative care in other surgical populations.

Despite growing evidence, there is a lack of comprehensive studies evaluating VR in the acute postoperative phase after lumbar disc surgery, particularly in comparison with conventional physical therapy protocols. This study aims to address this gap by investigating the effectiveness of VR-assisted physical therapy versus conventional physical therapy in patients undergoing lumbar discectomy.

The primary outcomes include pain intensity, pain threshold, and blood biomediator levels. Secondary outcomes include functional recovery, kinesiophobia, and anxiety. By systematically comparing both interventions, this trial seeks to determine the advantages and limitations of VR-assisted rehabilitation, with the goal of developing innovative, safe, and effective strategies for postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Undergoing lumbar discectomy surgery (L4-L5 or L5-S1 levels).
* Able to start postoperative physical therapy on day 1 after surgery.
* Willing and able to provide informed consent.
* Sufficient cognitive and physical ability to participate in physical therapy and virtual reality sessions.

Exclusion Criteria:

* History of previous lumbar spine surgery.
* Severe neurological deficits (e.g., cauda equina syndrome, progressive motor weakness).
* Diagnosed epilepsy, severe psychiatric illness, or other conditions contraindicate VR use.
* Significant visual or vestibular impairments preventing safe VR participation.
* Uncontrolled systemic diseases (e.g., cardiovascular, respiratory, or metabolic instability).
* Pregnancy.
* Inability to understand study instructions or complete outcome assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Pain severity will be assessed using a 10 cm Visual Analog Scale (VAS), where participants mark their perceived pain level ranging from 0 (no pain) to 10 (worst imaginable pain). Both resting pain and pain during the most difficult daily activity will be recorded.
Pain Pressure Threshold (Algometry) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Pressure pain thresholds will be measured using an algometer applied to quadratus lumborum, tibialis anterior, and iliopsoas muscles. This method provides an objective evaluation of pain sensitivity in targeted muscle groups.
Blood Biomediators (CRP, Cortisol, Leukocyte Count) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Blood samples will be collected to analyze inflammatory and stress-related biomarkers associated with postoperative pain. Routine venous blood collection (8-10 cc) will be performed, and analyses will be conducted in a central laboratory.

SECONDARY OUTCOMES:
Functional Capacity (Timed Up and Go Test) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Participants will be asked to rise from a chair, walk 3 meters, turn around, walk back, and sit down. The total time will be recorded in seconds as an indicator of mobility and functional performance.
Functional Capacity (10-Meter Walk Test) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Participants will walk a 10-meter distance at a comfortable but fast pace. The time will be recorded, and gait speed will be calculated.
Kinesiophobia (Tampa Scale of Kinesiophobia) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Fear of movement and reinjury will be measured using the validated Turkish version of the 17-item Tampa Scale of Kinesiophobia. Higher scores indicate greater movement-related fear.
Anxiety and Depression (Hospital Anxiety and Depression Scale, HADS) | Baseline (Postoperative Day 1, before intervention) and at postoperative day 2 (upon completion of the intervention).
  Psychological status will be evaluated with the Hospital Anxiety and Depression Scale, which includes separate subscales for anxiety (HADS-A) and depression (HADS-D).
Treatment Satisfaction (Global Perceived Effect, GPE Scale) | Post-operative day 2 (after intervention completion).
  Participants will rate their overall improvement after the intervention compared to their pre-treatment condition on a 7-point Likert scale, ranging from "completely recovered" to "worse than ever."
Virtual Reality Sickness Questionnaire (VRSQ) (VR group only) | Immediately before and after each VR session, approximately 30 minutes apart.
  Presence and severity of VR-related symptoms such as dizziness, nausea, or visual discomfort will be assessed using the validated Turkish version of the Virtual Reality Sickness Questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Ankara
  - Hacettepe University Hospital Neurosurgery Department, Ankara, Ankara

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because of patient privacy and confidentiality concerns.

REFERENCES:
- [Background] Avila L, da Silva MD, Neves ML, Abreu AR, Fiuza CR, Fukusawa L, de Sa Ferreira A, Meziat-Filho N. Effectiveness of Cognitive Functional Therapy Versus Core Exercises and Manual Therapy in Patients With Chronic Low Back Pain After Spinal Surgery: Randomized Controlled Trial. Phys Ther. 2024 Jan 1;104(1):pzad105. doi: 10.1093/ptj/pzad105. PMID 37548608
- [Background] He W, Wang Q, Hu J, Lin S, Zhang K, Wang F, Xu C, Li F, Xiao J, Li X, Tang F. A randomized trial on the application of a nurse-led early rehabilitation program after minimally invasive lumbar internal fixation. Ann Palliat Med. 2021 Sep;10(9):9820-9829. doi: 10.21037/apm-21-2294. PMID 34628908